CLINICAL TRIAL: NCT05258695
Title: American Orthopedic Foot and Ankle Society Hallux Metatarsophalangeal-interphalangeal Joint Scale (AOFAS Hallux MTP-IP)
Brief Title: The Turkish Version of the AOFAS Hallux MTP-IP
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 35
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2022-04

CONDITIONS: Foot Deformity; Hallux Deformity; Assessment, Self; Orthopedic Disorder
MeSH Terms: conditions — Foot Deformities; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The American Orthopedic Foot and Ankle Society hallux metatarsophalangeal-interphalangeal joint scale (AOFAS Hallux MTP-IP) is originally developed in English to evaluate the pain, function and alignment in patients with hallux deformities. The purpose of this study is to translate and cross-culturally adapt the AOFAS Hallux MTP-IP scale into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
The American Orthopedic Foot and Ankle Society hallux metatarsophalangeal-interphalangeal joint scale (AOFAS Hallux MTP-IP) is originally developed in English to evaluate joint function in patients with elbow stiffness. The purpose of this study is to translate and cross-culturally adapt the AOFAS Hallux MTP-IP scale into Turkish and investigate its psychometric properties. Approximately seventy patients with hallux deformities will be included. For cross-cultural adaptation, two bi-lingual translators will use the back-translation procedure. Within a 5-to-7-day period after the first assessment, the participants will complete the Turkish version of AOFAS Hallux MTP-IP (AOFAS Hallux MTP-IP-T) to evaluate test-retest reliability. Cronbach's alpha (α) will use to assess internal consistency. The correlation with the Turkish version of the Manchester-Oxford Foot Questionnaire (MOXFQ) and Short Form-12 will be determined to check the validity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Diagnosis of Hallux deformities
* Continuing follow-up and treatment in the orthopedic service
* Being able to follow simple instructions
* Being able to read and write in Turkish

Exclusion Criteria:

* Having any cardiovascular diseases, neurological disorders, rheumatic diseases, or psychiatric diseases
* Having peripheral nerve injury, peripheral neuropathy, or sensory loss in the lower extremity
* Having heterotopic ossification, myositis ossification, or post-traumatic ankylosing in the lower extremity
* Fracture, non-healing wound, or infection in the lower extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants are patients who have an hallux deformity and are treated in the orthopedic service. The participants with hallux deformity are directed for assessment following a confirmation by an orthopaedist based on the physical examinations and diagnostic imaging.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
The American Orthopedic Foot and Ankle Society hallux metatarsophalangeal-interphalangeal joint scale (AOFAS Hallux MTP-IP) | Day 1
  The American Orthopedic Foot and Ankle Society hallux metatarsophalangeal-interphalangeal joint scale (AOFAS Hallux MTP-IP) is composed of 9 items, distributed over 3 categories: pain (40 points), functional aspects (50 points), and alignment (10 points), for a total of 100 points.

SECONDARY OUTCOMES:
The American Orthopedic Foot and Ankle Society hallux metatarsophalangeal-interphalangeal joint scale (AOFAS Hallux MTP-IP) | Within a 5-to-7-day period after the first assessment (Day 1)
  The American Orthopedic Foot and Ankle Society hallux metatarsophalangeal-interphalangeal joint scale (AOFAS Hallux MTP-IP) is composed of 9 items, distributed over 3 categories: pain (40 points), functional aspects (50 points), and alignment (10 points), for a total of 100 points.
The Manchester-Oxford Foot Questionnaire (MOXFQ) | Day 1
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
Short Form-12 (SF-12) | Day 1
  Short Form-12 (SF-12), which is developed based on Short Form-36, consists of 12 items: 7 items dealing with the physical components scores (PCS-12) and 5 items related to the mental components scores (MCS-12) of SF-12.
  Range of both scores is 0 to 100, where the higher scores indicate better health related quality of life.
Visual Analogue Scale (VAS) | Day 1
  Pain intensity will be measured using the Visual Analogue Scale (VAS), in which the participants will be asked to indicate their perceived pain at rest, during activity, and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on a 10 cm line using a ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PhD, PT, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)